CLINICAL TRIAL: NCT07144501
Title: Prevalence of Liver Dysfunction in Paediatric Patients With Congenital Heart Disease: A Cross-Sectional Study at Assiut University Children Hospital.
Brief Title: Prevalence of Liver Dysfunction in Pediatric Patients With Congenital Heart Disease at Assiut.
Acronym: CHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Nassar Mohamed Ahmed, Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: YNMA22491; Assiut University (Other: Hospital of Faculty of Medicine at Assiut University)
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease; Liver Dysfunction
Keywords: CHD; Liver dysfunction
MeSH Terms: conditions — Heart Defects, Congenital; Liver Diseases | interventions — Ultrasonography; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHD patients (Experimental): A- Full History Taking:
  B- General Examination:
  C- Cardiac Examination:
  1. Physical examination
  2. Echocardiography
  D- Hepatic Examination:
  1. Physical examination
  2. Biochemical Markers: To assess hepatic function in congenital heart disease (CHD) patients, blood samples will be collected from all patients in our study
  3. Abdominal ultrasound:
  Interventions: Diagnostic Test: Ultrasonography; Procedure: Blood Sampling

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasound, also known as sonography or ultrasonography, is a medical imaging technique that uses high-frequency sound waves to create real-time images of internal body structures
Procedure: Blood Sampling — To assess hepatic function in congenital heart disease (CHD) patients, blood samples will be collected from all patients in our study for:
  * Alanine Transferase (ALT).
  * Aspartate Aminotransferase (AST).
  * Gamma Glutamyl Transferase (GGT).
  * Alkaline Phosphatase (ALP).
  * Total/direct bilirubin.
  * Albumin.
  * Prothrombin time.
  * International Normalized Ratio (INR).
  * Platelet count.

SUMMARY:
Liver dysfunction is a well-documented complication in patients with congenital heart disease (CHD). The mechanisms leading to hepatic dysfunction may be multifactorial. Key risk factors for liver dysfunction in CHD include prolonged hypoxemia, high venous pressure, and prolonged duration of heart disease.

While global studies have extensively explored this association, the prevalence of liver dysfunction in CHD varies, with studies reporting hepatic fibrosis in 30-40% of Fontan patients, while regional data, particularly from Egypt, remain limited.

In this research we aim to determine the prevalence of biochemical and radiological hepatic abnormalities in pediatric CHD patients attending Assiut University Children's Hospital.

DETAILED DESCRIPTION:
Liver dysfunction is a well-documented complication in patients with congenital heart disease (CHD), primarily due to chronic venous congestion, reduced cardiac output, and hypoxemia. The pathophysiology involves hepatic congestion secondary to right-sided heart failure, leading to fibrosis and cirrhosis in advanced cases. While global studies have extensively explored this association, regional data, particularly from Egypt, remain limited. In this research we aim to investigate liver dysfunction in CHD patients, with a specific focus on research conducted in Assiut, Egypt, to address gaps in localized clinical understanding.

Hepatic complications are common in patients with CHD, resulting either from the primary cardiac defect or from palliative surgical procedures performed in infancy or childhood or from transfusion- or drug-related hepatitis. Given that such patients increasingly require the expertise of a hepatologist. There are several known associations between primary liver disease and concomitant CHD defects such as Abernethy malformation, Alagille syndrome, and Biliary Atresia Splenic Malformation syndrome (BASM).

However, hepatic disease as a result of CHD is more common than cardiac disease associated with liver disease. In these cases, hepatic dysfunction may ensue as a result of the primary cardiac defect or as a result of surgical palliation, especially in patients with single-ventricle physiology (e.g., tricuspid atresia). The mechanisms leading to hepatic dysfunction may be multifactorial. As an example, hepatic dysfunction may result from a combination of passive venous congestion of the liver and hypoxia, with the latter being driven by the CHD or concomitant pulmonary disease. Volume overload and low cardiac output may lead to both congestive hepatopathy and hepatic ischemia.

Several factors may interact to lead to end-stage liver disease. For example, patients with underlying liver disease (e.g., viral hepatitis, alcohol, or obesity) may be more susceptible to liver injury as a result of decreased functional mass. In addition, the presence of cardiac disease and subsequent passive congestion may itself predispose the liver to hepatic injury. Hypoxemia in cyanotic CHD further aggravates hepatocellular damage, necessitating routine hepatic monitoring in this population.

Globally, the prevalence of liver dysfunction in CHD varies, with studies reporting hepatic fibrosis in 30-40% of Fontan patients. Data from developing regions, including Egypt, are scarce. A recent study highlighted elevated liver enzymes in CHD patients, emphasizing the role of delayed surgical intervention in disease progression. Such findings underscore the necessity for expanded research on hepatic complications in Egyptian CHD cohorts.

Key risk factors for liver dysfunction in CHD include prolonged hypoxemia, high venous pressure, and prolonged duration of heart disease. Cyanotic CHD patients exhibit higher hepatic injury markers compared to acyanotic counterparts. In Egypt, socioeconomic barriers often delay corrective surgeries, exacerbating hepatic damage. Early intervention and regular hepatic surveillance are critical to improving outcomes.

Despite global advancements, Egyptian studies on CHD-related liver dysfunction are limited. A 2016 Cairo University study identified a high prevalence of abnormal liver function tests among CHD patients but lacked longitudinal follow-up. Further research is needed to establish region-specific diagnostic and therapeutic protocols, considering local healthcare challenges.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pediatric CHD patients attending Assiut University Children's Hospital.
* Age: from birth up to 16 years old.

Exclusion Criteria:

* Patients with primary liver disease.
* Recent cardiac surgery (<3 m) (to exclude acute postoperative liver injury).
* Active systemic infection/sepsis (to avoid confounding liver enzyme elevations).

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of hepatic dysfunction among CHD | 5 months
  To assess the prevalence of hepatic dysfunction among CHD patients attending Assiut University Children's Hospital

SECONDARY OUTCOMES:
To classify hepatic dysfunction with CHD | 4 months
  To classify hepatic dysfunction with CHD using the APRI index into mild, moderate, and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Duaa Raafat, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University Children Hospital., Asyut, Assiut City, Egypt

IPD SHARING:
Plan to Share IPD: No
The policy of data confidentiality will be strictly followed with anonymous and secure data storage.

REFERENCES:
- [Background] Malatino LS, Fiore CE, Costa M, Calandra C, Petrone G, Cacciola S. Circadian rhythm of plasma tryptophan in clinically healthy subjects and patients with endogenous depression. Chronobiologia. 1982 Jan-Mar;9(1):13-20. PMID 7140474
- See also: relationship between Congenital heart disease and the liver — https://pubmed.ncbi.nlm.nih.gov/22383293/